CLINICAL TRIAL: NCT04533503
Title: Post-Market Clinical Evaluation of the Gentuity High-Frequency Optical Coherence Tomography Imaging System and Vis-Rx Micro-Imaging Catheter
Brief Title: Vis-Rx Post-Market Evaluation
Acronym: Vis-Rx PME
Status: Completed | Type: Observational
Sponsor: Gentuity, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 003175
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- HF-OCT imaging: Enrolled subjects who meet lesion-specific eligibility criteria and undergo HF-OCT imaging
  Interventions: Device: HF-OCT Imaging with the Vis-Rx Micro-Imaging Catheter

INTERVENTIONS:
Device: HF-OCT Imaging with the Vis-Rx Micro-Imaging Catheter — Intracoronary HF-OCT imaging of the target lesion(s) during the procedure.

SUMMARY:
Post-market clinical evaluation of the Gentuity High-Frequency Optical Coherence Tomography (HF-OCT) System and the Vis-Rx Micro-Imaging Catheter for use in Percutaneous Coronary Intervention (PCI) procedures.

DETAILED DESCRIPTION:
Prospective, single-arm, unblinded, multi-center, post-market clinical evaluation assessing the imaging capabilities of the Gentuity HF-OCT System and the Vis-Rx Micro-Imaging Catheter for use in PCI procedures. Objectives are to evaluate the clinical and technical performance in the target patient population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Willing and able to provide written informed consent to participate
* Transluminal interventional procedure for their coronary arteries

General Exclusion Criteria:

* Bacteremia or sepsis
* Major coagulation system abnormalities
* Severe hemodynamic instability or shock
* Acute renal failure
* Disqualified for Coronary Artery Bypass Graft (CABG) surgery
* Disqualified for PCI procedure
* Currently enrolled in another study to evaluate an investigational device or medication

Lesion-Specific Exclusion Criteria:

* Total occlusion
* Coronary artery spasm
* Large thrombus (visible under angiography)
* Any target vessel which has undergone a bypass procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the cardiac catheterization lab who are candidates for transluminal interventional procedures
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Clinical performance | Immediately after the procedure
  Operator evaluation of performance via Likert scale
Technical performance | Up to 3 months following the procedure
  Objective measurement of image clarity of the HF-OCT images by an independent core lab

SECONDARY OUTCOMES:
Complete pullbacks | Up to 3 months following the procedure
  Percentage of HF-OCT images with maximum clear image length

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of South Florida, Tampa, Florida
  - Baptist Health Lexington, Lexington, Kentucky
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No